CLINICAL TRIAL: NCT04855253
Title: Phase I/II Trial Using E7777 to Enhance Regulatory T-Cell Depletion Prior to CAR-T Therapy for Relapsed/Refractory Large B-Cell Lymphomas
Brief Title: Ph I/II Study of E7777 Prior to CAR-T for R/R LBCL
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Accrual met
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2020LS100; MT2020-27 (Other: University of Minnesota Masonic Cancer Center)
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: DLBCL; Diffuse Large B Cell Lymphoma; High-grade B-cell Lymphoma; DLBCL Arising From Follicular Lymphoma
Keywords: E7777; Axicabtagene; Lisocabtagene; Tisagenlecleucel
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — E7777 fusion protein; fludarabine; Cyclophosphamide; tisagenlecleucel; axicabtagene ciloleucel

STUDY DESIGN:
Intervention Model Description: The Phase I study consists of two components: dose finding to establish a maximum tolerated dose (MTD) of E7777 and a small extension component to provide an estimate of efficacy at the MTD.
  A single dose of E7777 is given on Day -7, two days prior to the start of lymphodepleting chemotherapy. Up to 3 dose levels will be tested. The MTD is determined by using the continual reassessment method (CRM). Enrollment begins with Dose Level 1 using a cohort of two patients. Twenty one (21) days after the 2nd patient's CAR-T cell infusion the next cohort of 2 patients are assigned to the most appropriate strategy based on updated toxicity probabilities corresponding to the desired maximum toxicity rate of ≤ 25% as determined by the study statistician (or designee). Enrollment continues in cohorts of 2 separated by a minimum of 28 days until 20 patients are enrolled or 10 sequential patients are enrolled at the same dose level. No intra-cohort staggering is required.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose level 1 : E7777 at 5 mcg/kg (Experimental): Single dose of E7777 given on Day -7 two days prior to the start of lymphodepleting chemotherapy
  Interventions: Drug: E7777; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Tisagenlecleucel; Drug: Axicabtagene Ciloleucel; Drug: Lisocabtagene Maraleucel Intravenous Suspension
- Dose level 1 : E7777 at 7 mcg/kg (Experimental): Single dose of E7777 given on Day -7 two days prior to the start of lymphodepleting chemotherapy
  Interventions: Drug: E7777; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Tisagenlecleucel; Drug: Axicabtagene Ciloleucel; Drug: Lisocabtagene Maraleucel Intravenous Suspension
- Dose level 1 : E7777 at 9 mcg/kg (Experimental): Single dose of E7777 given on Day -7 two days prior to the start of lymphodepleting chemotherapy
  Interventions: Drug: E7777; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Tisagenlecleucel; Drug: Axicabtagene Ciloleucel; Drug: Lisocabtagene Maraleucel Intravenous Suspension
- MTD from phase 1 (Experimental): Single dose of E7777 (Maximum tolerated dose level identified in phase 1) given on Day -7 two days prior to the start of lymphodepleting chemotherapy
  Interventions: Drug: E7777; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Tisagenlecleucel; Drug: Axicabtagene Ciloleucel; Drug: Lisocabtagene Maraleucel Intravenous Suspension

INTERVENTIONS:
Drug: E7777 — E7777 is a recombinant fusion toxin consisting of full-length human IL-2 fused to the catalytic domains of diphtheria toxin. E7777 is preferentially bound to and internalized by cells expressing the high affinity form (CD25+) of the IL-2 receptor.
Drug: Fludarabine — Fludarabine 25 mg/m2 IV daily for 3 days. Days -5, -4 and -3. Taken in combination with Cyclophosphamide
Drug: Cyclophosphamide — Cyclophosphamide 250 mg/m2 IV daily for 3 days starting with the first dose of fludarabine. Days -5, -4 and -3.
Drug: Tisagenlecleucel — Patient will receive one FDA approved CAR-T product - Tisagenlecleucel/Kymriah, Axicabtagene Ciloleucel/Yescarta, or lisocabtagene maraleucel/Breyanzi) for the treatment of relapsed/refractory diffuse large B-cell lymphoma
  Other Names: kymriah
Drug: Axicabtagene Ciloleucel — Patient will receive one FDA approved CAR-T product - Tisagenlecleucel/Kymriah, Axicabtagene Ciloleucel/Yescarta, or lisocabtagene maraleucel/Breyanzi) for the treatment of relapsed/refractory diffuse large B-cell lymphoma
  Other Names: Yescarta
Drug: Lisocabtagene Maraleucel Intravenous Suspension — Patient will receive one FDA approved CAR-T product - Tisagenlecleucel/Kymriah, Axicabtagene Ciloleucel/Yescarta, or lisocabtagene maraleucel/Breyanzi) for the treatment of relapsed/refractory diffuse large B-cell lymphoma
  Other Names: Breyanzi

SUMMARY:
This is a multicenter Phase I study to determine the maximum tolerated dose (MTD) of E7777 when given prior to cyclophosphamide/fludarabine (CY/Flu) lymphodepletion (LD) chemotherapy and an FDAapproved CAR-T product Tisagenlecleucel/Kymriah, Axicabtagene Ciloleucel/Yescarta, or lisocabtagene maraleucel/Breyanzi) for the treatment of relapsed/refractory diffuse large B-cell lymphoma (DLBCL) or follicular lymphoma grade 3 who are at a higher risk for failure of CAR-T therapy

DETAILED DESCRIPTION:
E7777 is a recombinant fusion toxin consisting of full-length human IL-2 fused to the catalytic domains of diphtheria toxin. This trial is designed to augment lymphodepletion prior to CAR-T cells by administration of a targeted immunotoxin against CD25-expressing T-cells. CD25 is expressed at high levels on Tregs but also on activated effector T cells. The use of the CAR-T cell product and associated apheresis and LD chemotherapy is considered standard of care (SOC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a relapse or refractory (r/r) B cell lymphoma, for which treatment with tisagenleucel (Kymriah), Axicabtagene (Yescarta) or Lisocabtagene Maraleucel (Breyanzi) is planned, including :
* diffuse large B-cell lymphoma (DLBCL) not otherwise specified,
* high grade B-cell lymphoma
* DLBCL arising from follicular lymphoma
* Primary mediastinal B cell lymphoma
* Follicular lymphoma grade 3B
* And considered at high risk for progression after CAR-T therapy by meeting one or more of the following factors:
* refractory to last line of therapy/remission of less than 12 months
* myc over expression >40% in any prior biopsy or bcl2/bcl6 and c-myc re-arrangement (double/triple hit)

  * 2 sites of extranodal disease
* IPI ≥ 3
* Elevated LDH at the time of relapse
* Has secured coverage for Kymriah, Yescarta,Breyanzi administration
* Age 18 years or older at the time of signing the consent
* ECOG Performance status of 0, 1, or 2
* Adequate bone marrow reserve (may be transfusion dependent)
* Adequate organ function at enrollment and within 14 days of planned E7777 treatment as defined in Section 4.1.7
* Hemodynamically stable and LVEF ≥ 50% confirmed by echocardiogram or MUGA

  * Grade 1 dyspnea (CTCAE v5) and SpO2 > 91% on room air
* Sexually active females of child-bearing potential and males with partners of child bearing potential must agree to use effective contraception during therapy
* Provides voluntary written consent prior to the performance of any research related activities.

Exclusion Criteria:

* Pregnant or breastfeeding - Females of childbearing potential must have a blood test or urine study within 14 days prior to study enrollment to rule out pregnancy. All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (i.e., bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing)
* Known bone marrow involvement, if history of bone marrow involvement must have a BM biopsy to rule-out current involvement
* Prior allogeneic transplant
* Ocular disease or complaints visual acuity impairment, color or shape distortion, or blurred vision - potential participants are required to have an ophthalmological examine as part of screening
* Active CNS involvement by malignancy (history of CNS disease with negative CSF by flow cytometry and/or stable findings on brain MRI are acceptable)
* Uncontrolled active hepatitis B or hepatitis C
* Active or inactive HIV infection
* Untreated active bacterial, viral or fungal infection (e.g. blood culture positive ≤ 72 hours prior to enrollment)
* History of heart failure or pulmonary edema, evidence of pleural effusion or active lower extremity edema
* Uncontrolled unstable angina and/or myocardial infarction within 3 months of enrollment
* Investigational medicinal product within the last 7 days prior to apheresis or CAR-T infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Establish maximum tolerated dose (MTD) | 1 month
  The primary objective of this Phase I study is to establish a maximum tolerated dose (MTD) of E7777 when given prior to standard of care CAR-T therapy product for the treatment of relapsed/refractory B-cell lymphoma who are at a higher risk for failure of CAR-T therapy.

SECONDARY OUTCOMES:
Number of participants experiencing adverse events | 100 days Post E7777 infusion
  Number of participants experiencing adverse events related to E7777 to determine safety of the E7777
Number of participants experiencing disease free survival (DFS) | 1 year Post E7777 infusion
  Number of participants experiencing disease free survival (DFS) at 1 year
Number of participants experiencing overall survival (OS) | 1 year Post E7777 infusion
  Number of participants experiencing overall survival (DFS) at 1 year
Number of non-relapse mortality incidents at day 100 | 100 days Post E7777 infusion
  Number of participants experiencing non-relapse mortality at day 100 post E7777 infusion
Number of Grade 3 or 4 cytokine release syndrome (CRS) incidents | 28 Days Post E7777 infusion
  Number of participants experiencing Grade 3 or 4 cytokine release syndrome (CRS) after CAR-T cell therapy.
Number of Grade 3 or 4 immune effector cell associated neurotoxicity (ICAN) syndrome incidents | 28 Days Post E7777 infusion
  Number of participants experiencing Grade 3 or 4 immune effector cell associated neurotoxicity (ICAN) syndrome after CAR-T cell therapy.
Number of participants experiencing dose limiting toxicity events | 28 Days Post E7777 infusion
  Dose Limiting Toxicity (DLT) is defined as any of the following events based on CTCAE v5 from the 1st infusion of E7777 through 21 days after the administration of CAR-T:
  * Grade 4 infusion related reaction (IRR) associated with E7777
  * Grade 4 or Grade 3 capillary leak syndrome (CLS)
  * Grade 3 or 4 liver function test abnormality that do not resolve to <Grade 2 within 5 days
  * Grade 3 or 4 non-hematologic toxicity event that occurs after the administration of E7777 and before lymphodepleting therapy
  * Any adverse event that results in a delay of lymphodepleting therapy for more than 72 hours and attributed to E7777
  * Any Grade 5 adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Veronika Bachanova, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota, Masonic Cancer Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Mahdi HS, Woodall-Jappe M, Singh P, Czuczman MS. Targeting regulatory T cells by E7777 enhances CD8 T-cell-mediated anti-tumor activity and extends survival benefit of anti-PD-1 in solid tumor models. Front Immunol. 2023 Oct 27;14:1268979. doi: 10.3389/fimmu.2023.1268979. eCollection 2023. PMID 38022532